CLINICAL TRIAL: NCT01748227
Title: Improving Pain Using Peer RE-inforced Self-management Skills (IMPPRESS)
Brief Title: IMproving Pain Using Peer RE-inforced Self-management Skills
Acronym: IMPPRESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: RRP 12-438
Record Dates: First submitted 2012-11-21; First posted 2012-12-12 (Estimated); Results first posted 2015-03-19 (Estimated); Last update posted 2015-05-15 (Estimated); Status verified 2015-04

CONDITIONS: Chronic Pain
Keywords: self-management; peer support; social support
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Peer-Coached Pain Self-Management (Other): Participants (n=20) were assigned to a peer coach, who delivered self-management instruction one-on-one over a 4-month period.
  Interventions: Behavioral: Peer-Delivered Pain Self-Management

INTERVENTIONS:
Behavioral: Peer-Delivered Pain Self-Management — Patients (n=20) were assigned a peer coach to meet with for 4 months to discuss pain self-management.

SUMMARY:
The overall purpose of this pilot study is to conduct a formative evaluation of (veteran)peer delivery of a chronic pain self-management program to veterans with chronic musculoskeletal pain.

Our specific aims are as follows:

Aim 1: Evaluate the feasibility of identifying, recruiting, training, and retaining veteran peers to implement a self-management program for chronic pain.

Aim 2: Identify facilitators and barriers to peer-delivery of a chronic pain self-management program.

Aim 3: Convene an expert panel to review the results of Aims 1 and 2, help to interpret the results, and plan next steps.

DETAILED DESCRIPTION:
This is a one-arm pilot study with a pretest/posttest design. Thus, participants' (n=20) baseline scores were compared to their final outcome assessment scores (i.e., change scores.) There was no control group.

This study is an intervention using peer coaches to deliver pain self-management instruction to patients. Peer coaches thus delivered the intervention and underwent a 3-hour training session prior to initiation of the study. Because peers served as intervention facilitators and not as recipients of the intervention, this study was not focused on peer outcomes.

Patients (n=20) attended a 2-hour didactic session led by the study nurse. Then patients were assigned a peer (2 patients per peer). Patients met with their peers for 4 months to discuss pain self-management with the guidance of a study manual. Peers were asked to contact patients a minimum of bi-weekly via telephone or in-person.

Peers reviewed each of the topic areas covered in the self-management manual. Peers reviewed a different topic each session, ask if the patient has questions, and discuss his or her personal experience with the topic being covered during that session. Modeling what the nurse care manager has done in prior studies, peers worked with patients to help them to set goals and to evaluate whether these goals are realistic. A new goal was set at each session, with the peer following up on the previous goals with the patient, whether they were accomplished, and if not, possible courses of action (e.g., modifying the goal or offering other advice to accomplish the goal). Throughout these sessions peers were encouraged to draw on their own experiences and how they personally overcame obstacles and handled setbacks and frustrations. Peers did not advise on or discuss medications or medical questions with patients.

Participating patients (n=20) were given outcome assessments at baseline and at 4-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Peers will be eligible if they have chronic musculoskeletal pain and have completed a pain self-management program from any of these chronic pain trials:

  * Stepped Care for Depression and Musculoskeletal Pain (SCAMP)
  * Evaluation of Stepped Care for Chronic Pain in Iraq and Afghanistan Veterans (ESCAPE)
  * CAre Management for the Effective use of Opioids (CAMEO)
  * Or participants of the VA Pain School or VA Pain program
  * Peers may also be recommended by their primary care providers at the VA
* Eligible patients must have musculoskeletal pain in the low back, cervical spine, or extremities (hip, knee, or shoulder) that has persisted for 3 months
* And have pain of at least moderate intensity as defined by a Brief Pain Inventory score 5

Exclusion Criteria:

* Patients will be excluded if they have active suicidal ideation
* Have been hospitalized for psychiatric or substance abuse reasons in the last 6 months pending back surgery
* Current substance dependence
* Severe medical conditions (e.g., New York Heart Association Class III or IV heart failure) that precludes participation
* Or severe hearing or speech impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-01; Primary Completion 2013-10 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Sassi Matthias, PhD MS BA, Principal Investigator — Richard L. Roudebush VA Medical Center, Indianapolis, IN
Locations (1):
- Richard L. Roudebush VA Medical Center, Indianapolis, IN, Indianapolis, Indiana, United States

REFERENCES:
- [Result] Matthias MS, McGuire AB, Kukla M, Daggy J, Myers LJ, Bair MJ. A brief peer support intervention for veterans with chronic musculoskeletal pain: a pilot study of feasibility and effectiveness. Pain Med. 2015 Jan;16(1):81-7. doi: 10.1111/pme.12571. Epub 2014 Oct 14. PMID 25312858
- [Result] Matthias MS, Kukla ME, McGuire AB, Bair MJ. Peer support for chronic pain self-management: A qualitative study of peer coaches' experiences. [Abstract]. Journal of general internal medicine. 2014 Apr 16; 29(1):169-170.
- [Result] Matthias MS, McGuire AB, Kukla ME, Daggy J, Myers L, Bair MJ. Effectiveness of a brief peer support intervention for veterans with chronic pain. [Abstract]. Journal of general internal medicine. 2014 Apr 16; 29(1):80.
- [Derived] Matthias MS, Kukla M, McGuire AB, Bair MJ. How Do Patients with Chronic Pain Benefit from a Peer-Supported Pain Self-Management Intervention? A Qualitative Investigation. Pain Med. 2016 Dec;17(12):2247-2255. doi: 10.1093/pm/pnw138. Epub 2016 Jul 8. PMID 28025359

RESULTS

PARTICIPANT FLOW:
Groups:
- Pain Self-Management: Training of (veteran) peers to deliver pain self-management materials to veterans with chronic pain
  Pain Self-Management: Training of veteran peers to deliver pain self-management material to veterans with chronic pain. Veteran peers will then be assigned 2 patients with chronic pain to work with over the next 4 months on pain self-management.
Period: Overall Study
Arm/Group | Pain Self-Management
Started | 20
Completed | 17
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Pain Self-Management
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 58 [35 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 17
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Pain/Enjoyment of Life/General Activity
Description: 3-item version of the Brief Pain Inventory. Possible range: 0-30. 0=no pain/interference, 30=maximum pain/interference. Thus lower values represent a better outcome.
Time Frame: Change from baseline to 4 month assessment
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Pain Self-Management: Peer delivery of pain self-management to veterans
  Trained peers were each assigned 2 veterans to meet with regularly for 4 months and discuss pain self-management and coping strategies.
Arm/Group | Pain Self-Management
Number analyzed (Participants) | 17
units on a scale | -1.24 (4.60)

2. Secondary Outcome: Pain Catastrophizing Scale
Description: Pain Catastrophizing Scale. 13-item scale. Possible score range 0-52, with lower scores representing improvement.
Time Frame: Baseline and 4 month assessment (final assessment)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pain Self-Management
Number analyzed (Participants) | 17
units on a scale | -5.12 (12.93)

3. Secondary Outcome: Multidimensional Perceived Social Support Scale (MPSS).
Description: 12 items, possible range 12-84 with higher scores indicating higher social support (i.e., better outcomes).
Time Frame: Baseline and 4 month for Statistical Package for Social Scientists (SPSS) and only 4 month final interview for Working Alliance
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pain Self-Management
Number analyzed (Participants) | 17
units on a scale | 6.96 (16.60)

4. Secondary Outcome: Patient Reported Outcome Measurement System (PROMIS)
Description: Possible scores range 0-100. Higher scores represent higher pain interference. Thus lower scores represent better outcomes.
Time Frame: Change from baseline to 4 month assessment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pain Self-Management
Number analyzed (Participants) | 17
units on a scale | -4.18 (11.39)

5. Secondary Outcome: Pain Centrality Scale
Description: Possible range 10-50. Higher scores indicate higher pain centrality, i.e., worse outcomes.
Time Frame: 4 month assessment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pain Self-Management
Number analyzed (Participants) | 17
units on a scale | -5.29 (8.79)

ADVERSE EVENTS:
Arm/Group | Pain Self-Management
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

LIMITATIONS AND CAVEATS:
This was a pilot study to examine feasibility and preliminary effectiveness of peer support for veterans with chronic pain. Because of the small sample size and pretest/posttest design of the study, results should be interpreted with caution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes